CLINICAL TRIAL: NCT06583213
Title: Comparative Study Between Conventional Spinal Anaesthesia and Fractional Spinal Anaesthesia on Systemic Haemodynamics in Frail Elderly Hip Fracture Patients
Brief Title: Conventional Spinal Anaesthesia Versus Fractional Spinal Anaesthesia on Hemodynamics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU MD76/2024
Record Dates: First submitted 2024-06-23; First posted 2024-09-03 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-05

CONDITIONS: Hip Fractures
Keywords: fractional spinal
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fractional Spinal Anaesthesia. Group A. (Experimental): An intrathecal catheter 20 G will be then inserted 4-5 cm into the intrathecal space.This technique of SA will be performed on all patients , the needle should be inserted between L3 and L4 space or L4 and L5 space in order to avoid injury to the spinal cord. An intrathecal mixture (5mL) containing 3 mg/ml hyperbaric bupivacaine and 1 μg/ml dexmedetomidine will be prepared. Intrathecal anaesthesia will be induced by giving 2 mL (6 mg of hyperbaric bupivacaine and 2 μg of dexmedetomidine ) of the mixture, followed by a second 2 mL injection after 25 min.
  Interventions: Procedure: Fractional Spinal Anaesthesia.; Procedure: Conventional Spinal Anaesthesia
- Conventional Spinal Anaesthesia. Group B. (Active Comparator): Intrathecal anaesthesia will be induced by giving 12.5 mg Hyperbaric bupivacaine (2.5mL) and 4 μg of dexmedetomidine (1mL) (i.e., a total intrathecal dose (3.5 mL) of 12.5mg of hyperbaric bupivacaine and 4 μg of dexmedetomidine ).
  Sensory level will be monitored by "cold spray". Haemodynamic recordings will be documented every five minutes up until 45 minutes.
  Interventions: Procedure: Fractional Spinal Anaesthesia.; Procedure: Conventional Spinal Anaesthesia

INTERVENTIONS:
Procedure: Fractional Spinal Anaesthesia. — An intrathecal catheter 20 G will be then inserted 4-5 cm into the intrathecal space.This technique of SA will be performed on all patients , the needle should be inserted between L3 and L4 space or L4 and L5 space in order to avoid injury to the spinal cord. An intrathecal mixture (5mL) containing 3 mg/ml hyperbaric bupivacaine and 1 μg/ml dexmedetomidine will be prepared. Intrathecal anaesthesia will be induced by giving 2 mL (6 mg of hyperbaric bupivacaine and 2 μg of dexmedetomidine ) of the mixture, followed by a second 2 mL injection after 25 min. (i.e., a total intrathecal dose (4mL) of 12 mg of hyperbaric bupivacaine and 4 μg of dexmedetomidine ).
Procedure: Conventional Spinal Anaesthesia — Intrathecal anaesthesia will be induced by giving 12.5 mg Hyperbaric bupivacaine (2.5mL) and 4 μg of dexmedetomidine (1mL) (i.e., a total intrathecal dose (3.5 mL) of 12.5mg of hyperbaric bupivacaine and 4 μg of dexmedetomidine ). (Mohamed T et al., 2017).
  Sensory level will be monitored by "cold spray". Haemodynamic recordings will be documented every five minutes up until 45 minutes.

SUMMARY:
compare the systemic haemodynamic response to fractional spinal anaesthesia versus conventional spinal anaesthesia , in a group of elderly and comorbid patients with hip fracture.

DETAILED DESCRIPTION:
Spinal anaesthesia affects sympathetic chain activity, leading to a reduction in vasomotor tone.It was found that the incidence of hypotension following single-shot spinal anaesthesia, has previously been described as being 28-69%. As a matter of fact, autonomic nervous system function plays a key role in the development of haemodynamic instability and intraoperative hypotension . Haemodynamic stability should be considered as a primary intraoperative target, since several findings suggest avoiding systemic pressure drops . It was found that hypotension is primarily related to the overall dose injected ; however, several other variables, including the volume, the type of the anaesthetics injected, different adjuvant agents, and pre- and intraoperative factors, may impact the haemodynamic effect of the SA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hip fractures.
* Patients age >60 years old.
* ASA ≤ 3.

Exclusion Criteria:

* Patients on anticoagulant medication.
* Planned for general anaesthesia .
* Patients had atrial fibrillation.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Is to measure blood pressure change intra-operative operative operative (2 hours) | 2 hours
  blood pressure monitoring

SECONDARY OUTCOMES:
Postoperative pain score for 24 hours | within 24 hours
  pain score using the Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: ahmed saudi, professor, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No